CLINICAL TRIAL: NCT06270511
Title: A Phase 1, 2-Part Study to Evaluate the Relative Bioavailability of and Food-Effect on Pharmacokinetics of Different Formulations of S-337395, and to Assess the Safety, Tolerability, and Pharmacokinetics Following Multiple Doses of S-337395 in Healthy Adult Participants
Brief Title: A Study to Investigate Different Formulations of S-337395 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2222T1412
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
Keywords: S-337395; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Masking Description: Part A will be open label; Part B will be double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Open Label (Experimental): Participants will receive different formulations of S-337395 without food and with food.
  Interventions: Drug: S-337395
- Part B: Double Blind (Experimental): Participants will receive S-337395 or placebo.
  Interventions: Drug: S-337395; Drug: Placebo

INTERVENTIONS:
Drug: S-337395 — Administered as an oral suspension.
Drug: Placebo — Administered as an oral suspension.
  Arms: Part B: Double Blind

SUMMARY:
The aim of this study is to investigate different formulations of S-337395.

DETAILED DESCRIPTION:
This single-center study comprises an open-label, randomized, crossover study, and a double-blinded, placebo-controlled, randomized, multiple-dose study to examine the relative bioavailability, food effect, pharmacokinetics, safety, and tolerability of different formulations of S-337395.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body mass index within the range of 18.5 to approximately 30.0 kilograms/meter squared (inclusive) at screening.
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for those participating in clinical studies.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the investigational intervention; or interfering with the interpretation of data.
* Lymphoma, leukemia, or any malignancy in the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Sensitivity to S-337395, or any components of the formulation, or drug or other allergy, that in the opinion of the investigator, contraindicates participation in the study.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Part A: Plasma Concentration of S-337395 | Days 1-5, 8-12, and 15-19 (Predose, up to 96 hours post dose)
Part B: Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 21

SECONDARY OUTCOMES:
Part A: Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 29
Part A: Plasma Concentration of S-337395 (Venous Samples Versus Capillary Microsamples) | Venous: Days 1-5, 8-12, and 15-19 (Predose, up to 96 hours post dose); Capillary: Days 1, 2, 8, and 9 (Up to 24 hours post dose)
Part B: Plasma Concentration of S-337395 | Days 1-12 (Predose, up to 96 hours post dose)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Lenexa, Lenexa, Kansas, United States